CLINICAL TRIAL: NCT01743989
Title: A Prospective, Randomized, Open Label, Two Arm Phase III Study to Evaluate Treatment Free Remission (TFR) Rate in Patients With Philadelphia-positive CML After Two Different Durations of Consolidation Treatment With Nilotinib 300mg BID.
Brief Title: A Randomized Phase III Study to Assess the Effect of a Longer Duration of Consolidation Treatment With Nilotinib on TFR in CP CML.
Acronym: ENESTPath
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AIC05; 2012-005124-15 (EudraCT Number)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Philadelphia Chromosome Positive (PH+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Keywords: Adult; Chronic myelogenous leukemia (CML); Chronic myeloid leukemia (CML); Chronic myelocytic leukemia (CML); Acute Lymphoblastic Leukemia (ALL) Philadelphia chromosome positive; Acute Lymphoid Leukemia; Suboptimal molecular response
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nilotinib

STUDY DESIGN:
Intervention Model Description: All participants received 24 months of study treatment. After 24 months of treatment, eligible participants (i.e. those deemed to have achieved sustained molecular response) were randomized to one of the two study arms on a continued open-label basis.
  Participants not achieving sustained molecular response after 24 months of treatment were not randomized but remained in the study until the 5-year study period was completed (Not randomized arm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nilotinib 24-month treatment (Experimental): Participants were treated with nilotinib 300mg BID for 24 months and, thereafter, entered the 36-month TFR phase
  Interventions: Drug: Nilotinib
- Nilotinib 36-month treatment (Experimental): Participants were treated with nilotinib 300mg BID for 36 months and, thereafter, entered the 24-month TFR phase
  Interventions: Drug: Nilotinib
- Not randomized (Experimental): Participants were treated with nolotinib 300mg BID for 24 months, but did not achieve a sustained molecular response after 24 months of treatment.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Participants received a daily oral nilotinib dose of 300 mg BID, given as two 150 mg capsules BID.
  Other Names: AMN107

SUMMARY:
This study aimed to assess the optimal duration of nilotinib 300 mg twice daily (BID) consolidation treatment in patients with Philadelphia chromosome-positive (Ph+) chronic myeloid leukemia (CML), in order that patients remained in treatment-free remission (≥MR4.0) without molecular relapse 12 months after starting the Treatment-Free Remission (TFR) phase.

DETAILED DESCRIPTION:
This was a prospective, randomized, open-label, multicenter Phase III study. The study design was made up of 3 phases:

* Nilotinib induction phase: 12 months
* Nilotinib consolidation phase: 12 or 24 months, depending on randomization
* Nilotinib treatment-free remission (TFR) phase: 24 or 36 months, depending on randomization.

Subjects were enrolled into the study and were treated with nilotinib 300mg twice daily (BID) for 24 months, during the induction (12 months) and consolidation (12 months) phases. At the end of the first 24 months of treatment, participants achieving a sustained molecular response (defined as ≥ MR4.0, in 4 out of 5 real-time quantitative polymerase chain reaction (RQ-PCR) assessments, including the last assessment, in the last 12 months) were randomized on a 1:1 basis to either:

1. suspend nilotinib treatment immediately and enter the TFR phase for 36 months (Nilotinib 24-month treatment arm), or
2. continue nilotinib treatment for a further 12 months (post-randomization consolidation phase), then suspend treatment and enter the TFR phase for 24 months (Nilotinib 36-month treatment arm).

Participants not achieving a sustained molecular response at 24 months from treatment start were not eligible for randomization and were treated at the discretion of the investigator according to standard practice. Information on survival, stem cell transplantation, and status of the patient's disease was collected until death or until 5 years from study entry, whichever came first. Additionally, for Nilotinib 36-month treatment arm, participants who did not achieve a sustained molecular response at 36 months from treatment start, discontinued from the study and were treated according to standard practice and followed up until death or until 5 years from study entry, whichever came first.

Participants relapsing during the TFR phase entered the nilotinib re-treatment phase of the study, and were re-treated with the same dose of nilotinib as they were on before the TFR phase. These patients remained on study until the completion of the 5-year study period unless prematurely withdrawn and discontinued from the study for any reason specified in the Protocol.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of chronic phase Ph+ CML
* Previous first-line treatment with imatinib for a minimum of 2 years;
* Patient in complete cytogenetic response;

Key Exclusion Criteria:

* Previous achievement of MR4.0 at study entry;
* Previous treatment with other target cells inhibitors other than imatinib;
* Patients with any history of detectable atypical Leukemia transcripts or patients with detectable atypical leukemia transcripts at screening;
* Previous anticancer agents for Chronic myeloid leukemia other than imatinib except for cytoreduction;
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol;
* History of other active malignancies within the 5 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively;
* Patients who have not recovered from prior surgery;
* Treatment with other investigational agents within 4 weeks of Day 1;
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug

Other inclusion/exclusion criteria might apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2013-04-15 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (179):
- Austria (5):
  - Novartis Investigative Site, Linz, Upper Austria
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Rankweil
  - Novartis Investigative Site, Salzburg
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Czechia (2):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
- Denmark (2):
  - Novartis Investigative Site, Holstebro
  - Novartis Investigative Site, Roskilde
- Novartis Investigative Site, HUS Helsinki, Finland
- France (25):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Le Mans, Cedex 09
  - Novartis Investigative Site, Paris, Cedex 10
  - Novartis Investigative Site, Caen, Cedex
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Chalon-sur-Saône
  - Novartis Investigative Site, Chambéry
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Dunkirk
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Pontoise
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Toulouse
- Germany (32):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Eisenach
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Georgsmarienhütte
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamm
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lütten Klein
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Westerstede
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Würzburg
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Italy (43):
  - Novartis Investigative Site, Alessandria, AL
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Livorno, LI
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Potenza, PZ
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Pagani, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Taranto, TA
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Treviso, TV
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Mirano, VE
  - Novartis Investigative Site, Venezia, VE
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
  - Novartis Investigative Site, Perugia
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Poland (8):
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (6):
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Iași
  - Novartis Investigative Site, Sibiu
  - Novartis Investigative Site, Timișoara
- Serbia (3):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Niš
  - Novartis Investigative Site, Novi Sad
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Martin
- Novartis Investigative Site, Ljubljana, Slovenia
- Spain (28):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, León, Castille and León
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Pontevedra, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Granollers
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Santa Cruz de Tenerife
  - Novartis Investigative Site, Zaragoza
- Novartis Investigative Site, Stockholm, Sweden
- United Kingdom (3):
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Borghi L, Rosti G, Maggi A, Breccia M, Di Bona E, Iurlo A, La Barba G, Sportoletti P, Albano F, Galimberti S, Rivellini F, Cambrin GR, Capodanno I, Cuneo A, Bonifacio M, Sica S, Arcaini L, Capochiani E, Minotto C, Ciceri F, Crugnola M, Di Caprio L, Supekar S, Elena C, Baccarani M, Vegni E. Perspectives and Emotional Experiences of Patients With Chronic Myeloid Leukemia During ENESTPath Clinical Trial and Treatment-Free Remission: Rationale and Protocol of the Italian Substudy. Front Oncol. 2021 May 26;11:638689. doi: 10.3389/fonc.2021.638689. eCollection 2021. PMID 34123791

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For one participant randomized to Nilotinib 36-month treatment arm, the informed consent was not obtained prior to any study specific procedure. This participant discontinued the study before entering the TFR phase.
Groups:
- Not Randomized: Participants were treated with nilotinib 300mg BID for 24 months, but did not achieve a sustained molecular response after 24 months of treatment and were not randomized.
Period: Treatment Phase
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Started | 120 | 119 | 381
Participants Who Signed Informed Consent (Participants for whom informed consent was obtained prior to any study specific procedure) | 120 | 118 | 381
Completed | 119 | 104 | 0
Not Completed | 1 | 15 | 381
Not completed — Unstable MR4.0 | 0 | 6 | 263
Not completed — Adverse Event | 0 | 4 | 67
Not completed — Withdrawal by Subject | 1 | 3 | 28
Not completed — Death | 0 | 1 | 3
Not completed — Abnormal laboratory value(s) | 0 | 0 | 3
Not completed — Protocol deviation | 0 | 0 | 3
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Abnormal test procedure result(s) | 0 | 0 | 1
Not completed — Administrative problems | 0 | 0 | 1
Not completed — New cancer (CML) therapy | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Patient non-compliance to treatment | 0 | 0 | 3
Not completed — Not randomized by mistake | 0 | 0 | 1
Not completed — Included by mistake | 0 | 0 | 1
Period: TFR Phase
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Started | 119 | 104 | 0
Completed | 37 | 36 | 0
Not Completed | 82 | 68 | 0
Not completed — Relapse (Loss of MMR/Confirmed loss of MR4.0) | 82 | 59 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Logistical problems | 0 | 2 | 0
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: Re-treatment Phase
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Started | 74 | 55 | 0
Completed | 58 | 46 | 0
Not Completed | 16 | 9 | 0
Not completed — Adverse Event | 8 | 4 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Administrative problems | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Unstable MR | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized | Total
Number analyzed (Participants) | 120 | 119 | 381 | 620
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 106 | 98 | 308 | 512
  >=65 years | 14 | 21 | 73 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 129 | 226
  Male | 72 | 70 | 252 | 394
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 114 | 112 | 355 | 581
  Black | 0 | 1 | 4 | 5
  Asian | 0 | 0 | 2 | 2
  Native American | 0 | 1 | 1 | 2
  North African descent | 1 | 0 | 1 | 2
  Unknown | 0 | 1 | 5 | 6
  Other | 5 | 4 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Remained in Treatment Free Remission (TFR) Without Molecular Relapse 12 Months After Entering the TFR Phase
Description: Number of participants who remained in TFR (≥molecular response (MR) 4.0) without molecular relapse 12 months after entering the TFR phase (without re-starting nilotinib therapy) divided by the number of participants who entered the TFR phase and multiplied by 100.
  Molecular relapse during TFR is defined as the loss of major molecular response (MMR), or the confirmed loss of MR4.0 (defined by 3 consecutive tests less than MR4.0 assessed at 3 consecutive visits during TFR phase). Participants dropping out early from the study during the TFR phase were considered as unsuccessful TFR.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MMR is defined as≥3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤0.1% BCR-ABL.
  MR4.0 is defined as either detectable disease≤0.01% BCR-ABL or undetectable disease in cDNA with≥10,000 ABL transcripts
Time Frame: 12 months after entering the TFR phase, which is after 36 months from study treatment start for Nilotinib 24-month treatment arm and after 48 months from study treatment start for Nilotinib 36-month treatment arm
Population: All enrolled subjects who entered the TFR phase
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment
Number analyzed (Participants) | 119 | 104
Percentage of participants | 31.9 [23.7 to 41.1] | 37.5 [28.2 to 47.5]
Statistical Analysis 1: Comparison: Nilotinib 24-month Treatment vs Nilotinib 36-month Treatment; Test type: Superiority; p = 0.383, Chi-squared

2. Secondary Outcome: Cumulative Incidence of MMR During the Pre-randomization Induction/Consolidation Phase Among Participants Without That Response at Study Entry
Description: Number of participants who were in MMR during pre-randomization induction/consolidation phase divided by the number of participants without that response at baseline and multiplied by 100.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MMR is defined as ≥3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤0.1% BCR-ABL.
Time Frame: From baseline up to 24 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure who did not reach MMR at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Number analyzed (Participants) | 23 | 16 | 98
Percentage of participants
  Up to 3 months after study treatment start (pre-randomization) | 69.6 [47.1 to 86.8] | 37.5 [15.2 to 64.6] | 29.6 [20.8 to 39.7]
  Up to 6 months after study treatment start (pre-randomization) | 100 [85.2 to 100.0] | 100.0 [79.4 to 100.0] | 64.3 [54.0 to 73.7]
  Up to 9 months after study treatment start (pre-randomization) | 100 [85.2 to 100.0] | 100.0 [79.4 to 100.0] | 71.4 [61.4 to 80.1]
  Up to 12 months after study treatment start (pre-randomization) | 100 [85.2 to 100.0] | 100.0 [79.4 to 100.0] | 77.6 [68.0 to 85.4]
  Up to 15 months after study treatment start (pre-randomization) | 100 [85.2 to 100.0] | 100.0 [79.4 to 100.0] | 80.6 [71.4 to 87.9]
  Up to 18 months after study treatment start (pre-randomization) | 100 [85.2 to 100.0] | 100.0 [79.4 to 100.0] | 82.7 [73.7 to 89.6]
  Up to 21 months after study treatment start (pre-randomization) | 100 [85.2 to 100.0] | 100.0 [79.4 to 100.0] | 85.7 [77.2 to 92.0]
  Up to 24 months after study treatment start (pre-randomization) | 100 [85.2 to 100.0] | 100.0 [79.4 to 100.0] | 86.7 [78.4 to 92.7]

3. Secondary Outcome: Cumulative Incidence of MMR During the Post-randomization Consolidation Phase Among Participants Without That Response at Study Entry
Description: Number of participants who were in MMR during post-randomization consolidation phase divided by the number of participants without that response at baseline and multiplied by 100. Post-randomization consolidation phase corresponded to the 12-month additional treatment (after randomization) for Nilotinib 36-month treatment arm.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MMR is defined as ≥3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤0.1% BCR-ABL.
Time Frame: From randomization (month 24 after study treatment start) up to 36 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure who did not reach MMR at baseline. Only participants randomized to Nilotinib 36-month treatment arm entered the post-randomization consolidation phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 36-month Treatment
Number analyzed (Participants) | 16
Percentage of participants
  Up to 27 months after study treatment start (post-randomization) | 100.0 [79.4 to 100.0]
  Up to 30 months after study treatment start (post-randomization) | 100.0 [79.4 to 100.0]
  Up to 33 months after study treatment start (post-randomization) | 100.0 [79.4 to 100.0]
  Up to 36 months after study treatment start (post-randomization) | 100.0 [79.4 to 100.0]

4. Secondary Outcome: Cumulative Incidence of MR4.0 During the Pre-randomization Induction/Consolidation Phase Among Participants Without That Response at Study Entry
Description: Number of participants who were in MR4.0 during the pre-randomization induction/consolidation phase divided by the number of participants without that response at baseline and multiplied by 100.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.0 is defined as either detectable disease ≤0.01% BCR-ABL IS or undetectable disease in cDNA with ≥10,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From baseline up to 24 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure who did not reach MR4.0 at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Number analyzed (Participants) | 92 | 94 | 357
Percentage of participants
  Up to 3 months after study treatment start (pre-randomization) | 48.9 [38.3 to 59.6] | 38.3 [28.5 to 48.9] | 12.9 [9.6 to 16.8]
  Up to 6 months after study treatment start (pre-randomization) | 85.9 [77.1 to 92.3] | 81.9 [72.6 to 89.1] | 26.6 [22.1 to 31.5]
  Up to 9 months after study treatment start (pre-randomization) | 94.6 [87.8 to 98.2] | 92.6 [85.3 to 97.0] | 34.5 [29.5 to 39.6]
  Up to 12 months after study treatment start (pre-randomization) | 96.7 [90.8 to 99.3] | 98.9 [94.2 to 100.0] | 39.2 [34.1 to 44.5]
  Up to 15 months after study treatment start (pre-randomization) | 100.0 [96.1 to 100.0] | 98.9 [94.2 to 100.0] | 42.0 [36.8 to 47.3]
  Up to 18 months after study treatment start (pre-randomization) | 100.0 [96.1 to 100.0] | 100.0 [96.2 to 100.0] | 45.1 [39.9 to 50.4]
  Up to 21 months after study treatment start (pre-randomization) | 100.0 [96.1 to 100.0] | 100.0 [96.2 to 100.0] | 48.7 [43.4 to 54.1]
  Up to 24 months after study treatment start (pre-randomization) | 100.0 [96.1 to 100.0] | 100.0 [96.2 to 100.0] | 52.1 [46.8 to 57.4]

5. Secondary Outcome: Cumulative Incidence of MR4.0 During the Post-randomization Consolidation Phase Among Participants Without That Response at Study Entry
Description: Number of participants who were in MR4.0 during the post-randomization consolidation phase divided by the number of participants without that response at baseline and multiplied by 100. Post-randomization consolidation phase corresponded to the 12-month additional treatment (after randomization) for Nilotinib 36-month treatment arm.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.0 is defined as either detectable disease ≤0.01% BCR-ABL IS or undetectable disease in cDNA with ≥10,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From randomization (month 24 after study treatment start) up to 36 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure who did not reach MR4.0 at baseline. Only participants randomized to Nilotinib 36-month treatment arm entered the post-randomization consolidation phase
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 36-month Treatment
Number analyzed (Participants) | 94
Percentage of participants
  Up to 27 months after study treatment start (post-randomization) | 97.9 [92.5 to 99.7]
  Up to 30 months after study treatment start (post-randomization) | 97.9 [92.5 to 99.7]
  Up to 33 months after study treatment start (post-randomization) | 97.9 [92.5 to 99.7]
  Up to 36 months after study treatment start (post-randomization) | 97.9 [92.5 to 99.7]

6. Secondary Outcome: Cumulative Incidence of MR4.5 During the Pre-randomization Induction/Consolidation Phase Among Participants Without That Response at Study Entry
Description: Number of participants who were in MR4.5 during the pre-randomization induction/consolidation phase divided by the number of participants without that response at baseline and multiplied by 100.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.5 is defined as either detectable disease ≤ 0.0032% BCR-ABL IS; or undetectable disease within cDNA with ≥ 32,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From baseline up to 24 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure who did not reach MR4.5 at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Number analyzed (Participants) | 109 | 109 | 374
Percentage of participants
  Up to 3 months after study treatment start (pre-randomization) | 21.1 [13.9 to 30.0] | 17.4 [10.8 to 25.9] | 4.0 [2.3 to 6.5]
  Up to 6 months after study treatment start (pre-randomization) | 38.5 [29.4 to 48.3] | 38.5 [29.4 to 48.3] | 8.6 [5.9 to 11.9]
  Up to 9 months after study treatment start (pre-randomization) | 57.8 [48.0 to 67.2] | 54.1 [44.3 to 63.7] | 10.7 [7.8 to 14.3]
  Up to 12 months after study treatment start (pre-randomization) | 70.6 [61.2 to 79.0] | 65.1 [55.4 to 74.0] | 14.2 [10.8 to 18.1]
  Up to 15 months after study treatment start (pre-randomization) | 79.8 [71.1 to 86.9] | 76.1 [67.0 to 83.8] | 15.2 [11.8 to 19.3]
  Up to 18 months after study treatment start (pre-randomization) | 83.5 [75.2 to 89.9] | 80.7 [72.1 to 87.7] | 16.6 [13.0 to 20.7]
  Up to 21 months after study treatment start (pre-randomization) | 85.3 [77.3 to 91.4] | 84.4 [76.2 to 90.6] | 18.4 [14.7 to 22.8]
  Up to 24 months after study treatment start (pre-randomization) | 89.0 [81.6 to 94.2] | 89.0 [81.6 to 94.2] | 20.3 [16.4 to 24.8]

7. Secondary Outcome: Cumulative Incidence of MR4.5 During the Post-randomization Consolidation Phase Among Participants Without That Response at Study Entry
Description: Number of participants who were in MR4.5 during the post-randomization consolidation phase divided by the number of participants without that response at baseline and multiplied by 100. Post-randomization consolidation phase corresponded to the 12-month additional treatment (after randomization) for Nilotinib 36-month treatment arm.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.5 is defined as either detectable disease ≤ 0.0032% BCR-ABL IS; or undetectable disease within cDNA with ≥ 32,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From randomization (month 24 after study treatment start) up to 36 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure who did not reach MR4.5 at baseline. Only participants randomized to Nilotinib 36-month treatment arm entered the post-randomization consolidation phase
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 36-month Treatment
Number analyzed (Participants) | 109
Percentage of participants
  Up to 27 months after study treatment start (post-randomization) | 70.6 [61.2 to 79.0]
  Up to 30 months after study treatment start (post-randomization) | 76.1 [67.0 to 83.8]
  Up to 33 months after study treatment start (post-randomization) | 84.4 [76.2 to 90.6]
  Up to 36 months after study treatment start (post-randomization) | 87.2 [79.4 to 92.8]

8. Secondary Outcome: Cumulative Incidence of MMR During the Pre-randomization Induction/Consolidation Phase
Description: Number of participants who were in MMR during the pre-randomization induction/consolidation phase divided by the number of enrolled participants and multiplied by 100.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MMR is defined as ≥3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤0.1% BCR-ABL.
Time Frame: From baseline up to 24 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Number analyzed (Participants) | 120 | 118 | 381
Percentage of participants
  Baseline | 80.8 [72.6 to 87.4] | 86.4 [78.9 to 92.1] | 74.3 [69.6 to 78.6]
  Up to 3 months after study treatment start (pre-randomization) | 94.2 [88.4 to 97.6] | 91.5 [85.0 to 95.9] | 81.9 [77.7 to 85.6]
  Up to 6 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 90.8 [87.5 to 93.5]
  Up to 9 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 92.7 [89.6 to 95.1]
  Up to 12 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 94.2 [91.4 to 96.4]
  Up to 15 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 95.0 [92.3 to 97.0]
  Up to 18 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 95.5 [93.0 to 97.4]
  Up to 21 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 96.3 [93.9 to 98.0]
  Up to 24 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 96.6 [94.2 to 98.2]

9. Secondary Outcome: Cumulative Incidence of MMR During the Post-randomization Consolidation Phase
Description: Number of participants who were in MMR during the post-randomization consolidation phase divided by the number of enrolled participants and multiplied by 100. Post-randomization consolidation phase corresponded to the 12-month additional treatment (after randomization) for Nilotinib 36-month treatment arm.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MMR is defined as ≥3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤0.1% BCR-ABL.
Time Frame: From randomization (month 24 after study treatment start) up to 36 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure. Only participants randomized to Nilotinib 36-month treatment arm entered the post-randomization consolidation phase
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 36-month Treatment
Number analyzed (Participants) | 118
Percentage of participants
  Up to 27 months after study treatment start (post-randomization) | 98.3 [94.0 to 99.8]
  Up to 30 months after study treatment start (post-randomization) | 98.3 [94.0 to 99.8]
  Up to 33 months after study treatment start (post-randomization) | 98.3 [94.0 to 99.8]
  Up to 36 months after study treatment start (post-randomization) | 98.3 [94.0 to 99.8]

10. Secondary Outcome: Cumulative Incidence of MR4.0 During the Pre-randomization Induction/Consolidation Phase
Description: Number of participants who were in MR4.0 during the pre-randomization induction/consolidation phase divided by the number of enrolled participants and multiplied by 100.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.0 is defined as either detectable disease ≤0.01% BCR-ABL IS or undetectable disease in cDNA with ≥10,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From baseline up to 24 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Number analyzed (Participants) | 120 | 118 | 381
Percentage of participants
  Baseline | 23.3 [16.1 to 31.9] | 20.3 [13.5 to 28.7] | 6.3 [4.1 to 9.2]
  Up to 3 months after study treatment start (pre-randomization) | 60.8 [51.5 to 69.6] | 50.8 [41.5 to 60.2] | 18.4 [14.6 to 22.6]
  Up to 6 months after study treatment start (pre-randomization) | 89.2 [82.2 to 94.1] | 85.6 [77.9 to 91.4] | 31.2 [26.6 to 36.2]
  Up to 9 months after study treatment start (pre-randomization) | 95.8 [90.5 to 98.6] | 94.1 [88.2 to 97.6] | 38.6 [33.7 to 43.7]
  Up to 12 months after study treatment start (pre-randomization) | 97.5 [92.9 to 99.5] | 99.2 [95.4 to 100.0] | 43.0 [38.0 to 48.2]
  Up to 15 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 99.2 [95.4 to 100.0] | 45.7 [40.6 to 50.8]
  Up to 18 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 48.6 [43.4 to 53.7]
  Up to 21 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 52.0 [46.8 to 57.1]
  Up to 24 months after study treatment start (pre-randomization) | 100.0 [97.0 to 100.0] | 100.0 [96.9 to 100.0] | 55.1 [50.0 to 60.2]

11. Secondary Outcome: Cumulative Incidence of MR4.0 During the Post-randomization Consolidation Phase
Description: Number of participants who were in MR4.0 during the post-randomization consolidation phase divided by the number of enrolled participants and multiplied by 100. Post-randomization consolidation phase corresponded to the 12-month additional treatment (after randomization) for Nilotinib 36-month treatment arm.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.0 is defined as either detectable disease ≤0.01% BCR-ABL IS or undetectable disease in cDNA with ≥10,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From randomization (month 24 after study treatment start) up to 36 months after study treatment start
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 36-month Treatment
Number analyzed (Participants) | 118
Percentage of participants
  Up to 27 months after study treatment start (post-randomization) | 98.3 [94.0 to 99.8]
  Up to 30 months after study treatment start (post-randomization) | 98.3 [94.0 to 99.8]
  Up to 33 months after study treatment start (post-randomization) | 98.3 [94.0 to 99.8]
  Up to 36 months after study treatment start (post-randomization) | 98.3 [94.0 to 99.8]

12. Secondary Outcome: Cumulative Incidence of MR4.5 During the Pre-randomization Induction/Consolidation Phase
Description: Number of participants who were in MR4.5 during the pre-randomization induction/consolidation phase divided by the number of enrolled participants and multiplied by 100.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.5 is defined as either detectable disease ≤ 0.0032% BCR-ABL IS; or undetectable disease within cDNA with ≥ 32,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From baseline up to 24 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained before any study specific procedure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Number analyzed (Participants) | 120 | 118 | 381
Percentage of participants
  Baseline | 9.2 [4.7 to 15.8] | 7.6 [3.6 to 14.0] | 1.8 [0.7 to 3.8]
  Up to 3 months after study treatment start (pre-randomization) | 28.3 [20.5 to 37.3] | 23.7 [16.4 to 32.4] | 5.8 [3.7 to 8.6]
  Up to 6 months after study treatment start (pre-randomization) | 44.2 [35.1 to 53.5] | 43.2 [34.1 to 52.7] | 10.2 [7.4 to 13.7]
  Up to 9 months after study treatment start (pre-randomization) | 61.7 [52.4 to 70.4] | 57.6 [48.2 to 66.7] | 12.3 [9.2 to 16.1]
  Up to 12 months after study treatment start (pre-randomization) | 73.3 [64.5 to 81.0] | 67.8 [58.6 to 76.1] | 15.7 [12.2 to 19.8]
  Up to 15 months after study treatment start (pre-randomization) | 81.7 [73.6 to 88.1] | 78.0 [69.4 to 85.1] | 16.8 [13.2 to 20.9]
  Up to 18 months after study treatment start (pre-randomization) | 85.0 [77.3 to 90.9] | 82.2 [74.1 to 88.6] | 18.1 [14.4 to 22.4]
  Up to 21 months after study treatment start (pre-randomization) | 86.7 [79.3 to 92.2] | 85.6 [77.9 to 91.4] | 19.9 [16.1 to 24.3]
  Up to 24 months after study treatment start (pre-randomization) | 90.0 [83.2 to 94.7] | 89.8 [82.9 to 94.6] | 21.8 [17.7 to 26.3]

13. Secondary Outcome: Cumulative Incidence of MR4.5 During the Post-randomization Consolidation Phase
Description: Number of participants who were in MR4.5 during the post-randomization consolidation phase divided by the number of enrolled participants and multiplied by 100. Post-randomization consolidation phase corresponded to the 12-month additional treatment (after randomization) for Nilotinib 36-month treatment arm.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.5 is defined as either detectable disease ≤ 0.0032% BCR-ABL IS; or undetectable disease within cDNA with ≥ 32,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From randomization (month 24 after study treatment start) up to 36 months after study treatment start
Population: All enrolled subjects for whom written informed consent was obtained before any study specific procedure. Only participants randomized to Nilotinib 36-month treatment arm entered the post-randomization consolidation phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 36-month Treatment
Number analyzed (Participants) | 118
Percentage of participants
  Up to 27 months after study treatment start (post-randomization) | 72.9 [63.9 to 80.7]
  Up to 30 months after study treatment start (post-randomization) | 78.0 [69.4 to 85.1]
  Up to 33 months after study treatment start (post-randomization) | 85.6 [77.9 to 91.4]
  Up to 36 months after study treatment start (post-randomization) | 88.1 [80.9 to 93.4]

14. Secondary Outcome: Percentage of Participants Who Were in MMR During TFR Phase
Description: Number of participants who were in MMR at selected timepoints divided by the number of participants in the TFR phase and multiplied by 100. Participants randomized in Nilotinib 36-month treatment arm had a maximum of 24 months of TFR phase, whereas participants randomized in Nilotinib 24-month treatment arm had a maximum of 36 months of TFR phase.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MMR is defined as ≥3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤0.1% BCR-ABL.
Time Frame: From Month 1 after entering TFR phase up to 24 months after entering TFR phase for Nilotinib 36-month treatment arm and up to 36 months after entering TFR phase for Nilotinib 24-month treatment arm
Population: All enrolled subjects who entered the TFR phase
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment
Number analyzed (Participants) | 119 | 104
Percentage of participants
  Month 1 after entering TFR phase | 97.5 [92.8 to 99.5] | 94.2 [87.9 to 97.9]
  Month 2 after entering TFR phase | 84.9 [77.2 to 90.8] | 80.8 [71.9 to 87.8]
  Month 3 after entering TFR phase | 62.2 [52.8 to 70.9] | 61.5 [51.5 to 70.9]
  Month 4 after entering TFR phase | 51.3 [41.9 to 60.5] | 53.8 [43.8 to 63.7]
  Month 5 after entering TFR phase | 45.4 [36.2 to 54.8] | 46.2 [36.3 to 56.2]
  Month 6 after entering TFR phase | 42.9 [33.8 to 52.3] | 43.3 [33.6 to 53.4]
  Month 8 after entering TFR phase | 40.3 [31.5 to 49.7] | 43.3 [33.6 to 53.4]
  Month 10 after entering TFR phase | 38.7 [29.9 to 48.0] | 42.3 [32.7 to 52.4]
  Month 12 after entering TFR phase | 36.1 [27.5 to 45.5] | 39.4 [30.0 to 49.5]
  Month 15 after entering TFR phase | 35.3 [26.8 to 44.6] | 39.4 [30.0 to 49.5]
  Month 18 after entering TFR phase | 35.3 [26.8 to 44.6] | 39.4 [30.0 to 49.5]
  Month 21 after entering TFR phase | 34.5 [26.0 to 43.7] | 38.5 [29.1 to 48.5]
  Month 24 after entering TFR phase | 31.9 [23.7 to 41.1] | 35.6 [26.4 to 45.6]
  Month 27 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 27 after entering TFR phase | 31.9 [23.7 to 41.1] |
  Month 30 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 30 after entering TFR phase | 31.9 [23.7 to 41.1] |
  Month 33 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 33 after entering TFR phase | 30.3 [22.2 to 39.4] |
  Month 36 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 36 after entering TFR phase | 23.5 [16.2 to 32.2] |

15. Secondary Outcome: Percentage of Participants Who Were in MR4.0 During the TFR Phase
Description: Number of participants who were in MR4.0 at selected timepoints divided by the number of participants in the TFR phase and multiplied by 100. Participants randomized in Nilotinib 36-month treatment arm had a maximum of 24 months of TFR phase, whereas participants randomized in Nilotinib 24-month treatment arm had a maximum of 36 months of TFR phase.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.0 is defined as either detectable disease ≤0.01% BCR-ABL IS or undetectable disease in cDNA with ≥10,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From Month 1 after entering TFR phase up to 24 months after entering TFR phase for Nilotininb 36-months treatment arm and up to 36 months after entering TFR phase for Nilotinib 24-months treatment arm
Population: All enrolled subjects who entered the TFR phase
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Nilotinib 36-month Treatment Arm: Participants were treated with nilotinib 300mg BID for 36 months and, thereafter, entered the 24-month TFR phase
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment Arm
Number analyzed (Participants) | 119 | 104
Percentage of participants
  Month 1 after entering TFR phase | 87.4 [80.1 to 92.8] | 83.7 [75.1 to 90.2]
  Month 2 after entering TFR phase | 58.0 [48.6 to 67.0] | 56.7 [46.7 to 66.4]
  Month 3 after entering TFR phase | 39.5 [30.7 to 48.9] | 42.3 [32.7 to 52.4]
  Month 4 after entering TFR phase | 36.1 [27.5 to 45.5] | 42.3 [32.7 to 52.4]
  Month 5 after entering TFR phase | 32.8 [24.5 to 42.0] | 41.3 [31.8 to 51.4]
  Month 6 after entering TFR phase | 33.6 [25.2 to 42.9] | 38.5 [29.1 to 48.5]
  Month 8 after entering TFR phase | 34.5 [26.0 to 43.7] | 40.4 [30.9 to 50.5]
  Month 10 after entering TFR phase | 35.3 [26.8 to 44.6] | 38.5 [29.1 to 48.5]
  Month 12 after entering TFR phase | 31.9 [23.7 to 41.1] | 37.5 [28.2 to 47.5]
  Month 15 after entering TFR phase | 34.5 [26.0 to 43.7] | 34.6 [25.6 to 44.6]
  Month 18 after entering TFR phase | 33.6 [25.2 to 42.9] | 38.5 [29.1 to 48.5]
  Month 21 after entering TFR phase | 30.3 [22.2 to 39.4] | 32.7 [23.8 to 42.6]
  Month 24 after entering TFR phase | 29.4 [21.4 to 38.5] | 30.8 [22.1 to 40.6]
  Month 27 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 27 after entering TFR phase | 31.1 [22.9 to 40.2] |
  Month 30 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 30 after entering TFR phase | 30.3 [22.2 to 39.4] |
  Month 33 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 33 after entering TFR phase | 27.7 [19.9 to 36.7] |
  Month 36 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 36 after entering TFR phase | 26.1 [18.4 to 34.9] |

16. Secondary Outcome: Percentage of Participants Who Were in MR4.5 During the TFR Phase
Description: Number of participants who were in MR4.5 at selected timepoints divided by the number of participants in the TFR phase and multiplied by 100. Participants randomized in Nilotinib 36-month treatment arm had a maximum of 24 months of TFR phase, whereas participants randomized in Nilotinib 24-month treatment arm had a maximum of 36 months of TFR phase.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method. MR4.5 is defined as either detectable disease ≤ 0.0032% BCR-ABL IS; or undetectable disease within cDNA with ≥ 32,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From Month 1 after entering TFR phase up to 24 months after entering TFR phase for Nilotininb 36-month treatment arm and up to 36 months after entering TFR phase for Nilotinib 24-month treatment arm
Population: All enrolled subjects who entered the TFR phase
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment Arm
Number analyzed (Participants) | 119 | 104
Percentage of participants
  Month 3 after entering TFR phase | 21.8 [14.8 to 30.4] | 26.9 [18.7 to 36.5]
  Month 6 after entering TFR phase | 17.6 [11.3 to 25.7] | 28.8 [20.4 to 38.6]
  Month 12 after entering TFR phase | 20.2 [13.4 to 28.5] | 26.9 [18.7 to 36.5]
  Month 15 after entering TFR phase | 18.5 [12.0 to 26.6] | 23.1 [15.4 to 32.4]
  Month 18 after entering TFR phase | 25.2 [17.7 to 34.0] | 26.9 [18.7 to 36.5]
  Month 21 after entering TFR phase | 22.7 [15.5 to 31.3] | 22.1 [14.6 to 31.3]
  Month 24 after entering TFR phase | 24.4 [17.0 to 33.1] | 20.2 [13.0 to 29.2]
  Month 27 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 27 after entering TFR phase | 21.8 [14.8 to 30.4] |
  Month 30 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 30 after entering TFR phase | 22.7 [15.5 to 31.3] |
  Month 33 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 33 after entering TFR phase | 19.3 [12.7 to 27.6] |
  Month 36 after entering TFR phase: number analyzed (Participants) | 119 | 0
  Month 36 after entering TFR phase | 16.8 [10.6 to 24.8] |

17. Secondary Outcome: BCR-ABL Ratio (Expressed as a Percentage) During the Induction/Consolidation Phase
Description: BCR-ABL transcript ratio by international scale (IS) (expressed as a percentage) during the induction/consolidation phase. Participants randomized to Nilotinib 36-month treatment arm had 12-month additional consolidation phase (post-randomization).
Time Frame: From baseline up to 24 months after study treatment start for Nilotinib 24-month treatment arm and Not randomized participants; and up to 36 months after study treatment start for Nilotinib 36-month treatment arm.
Population: All enrolled subjects for whom written informed consent was obtained prior to any study specific procedure. Number analyzed signified number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment Arm | Not Randomized
Number analyzed (Participants) | 120 | 118 | 381
Percentage
  Baseline: number analyzed (Participants) | 120 | 117 | 380
  Baseline | 0.1367 (0.55144) | 0.0633 (0.12790) | 0.5509 (3.94256)
  Month 3 after study treatment start (pre-randomization): number analyzed (Participants) | 117 | 117 | 343
  Month 3 after study treatment start (pre-randomization) | 0.0106 (0.02660) | 0.0086 (0.01155) | 0.0728 (0.22537)
  Month 6 after study treatment start (pre-randomization): number analyzed (Participants) | 118 | 115 | 327
  Month 6 after study treatment start (pre-randomization) | 0.0052 (0.00631) | 0.0124 (0.05508) | 0.0530 (0.09587)
  Month 9 after study treatment start (pre-randomization): number analyzed (Participants) | 116 | 117 | 312
  Month 9 after study treatment start (pre-randomization) | 0.0049 (0.00809) | 0.0046 (0.00544) | 0.0573 (0.13905)
  Month 12 after study treatment start (pre-randomization): number analyzed (Participants) | 117 | 117 | 298
  Month 12 after study treatment start (pre-randomization) | 0.0044 (0.00611) | 0.0037 (0.00440) | 0.0772 (0.56398)
  Month 15 after study treatment start (pre-randomization): number analyzed (Participants) | 117 | 116 | 286
  Month 15 after study treatment start (pre-randomization) | 0.0035 (0.00591) | 0.0034 (0.00389) | 0.0669 (0.37209)
  Month 18 after study treatment start (pre-randomization): number analyzed (Participants) | 117 | 115 | 269
  Month 18 after study treatment start (pre-randomization) | 0.0029 (0.00354) | 0.0034 (0.00409) | 0.0462 (0.12284)
  Month 21 after study treatment start (pre-randomization): number analyzed (Participants) | 115 | 114 | 246
  Month 21 after study treatment start (pre-randomization) | 0.0028 (0.00319) | 0.0031 (0.00288) | 0.0390 (0.08271)
  Month 24 after study treatment start (pre-randomization): number analyzed (Participants) | 113 | 113 | 153
  Month 24 after study treatment start (pre-randomization) | 0.0027 (0.00424) | 0.0029 (0.00319) | 0.0325 (0.05140)
  Month 27 after study treatment start (post-randomization): number analyzed (Participants) | 0 | 112 | 0
  Month 27 after study treatment start (post-randomization) |  | 0.0089 (0.06119) |
  Month 30 after study treatment start (post-randomization): number analyzed (Participants) | 0 | 112 | 0
  Month 30 after study treatment start (post-randomization) |  | 0.0111 (0.08672) |
  Month 33 after study treatment start (post-randomization): number analyzed (Participants) | 0 | 111 | 0
  Month 33 after study treatment start (post-randomization) |  | 0.0025 (0.00439) |
  Month 36 after study treatment start (post-randomization): number analyzed (Participants) | 0 | 103 | 0
  Month 36 after study treatment start (post-randomization) |  | 0.0025 (0.00338) |

18. Secondary Outcome: BCR-ABL Ratio (Expressed as a Percentage) During the TFR Phase
Description: BCR-ABL/control gene (ABL) transcript ratio by international scale (IS) (expressed as a percentage) during the TFR phase. BCR-ABL is the fusion gene from breakpoint cluster region and Abelson genes.
  Participants randomized in Nilotinib 36-month treatment arm had a maximum of 24 months of TFR phase, whereas participants randomized in Nilotinib 24-month treatment arm had a maximum of 36 months of TFR phase.
Time Frame: as for outcome 14
Population: All enrolled subjects who entered the TFR phase. Number analyzed signified number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment Arm
Number analyzed (Participants) | 119 | 104
Percentage
  Month 1 after entering the TFR phase: number analyzed (Participants) | 116 | 99
  Month 1 after entering the TFR phase | 0.0042 (0.00621) | 0.0074 (0.02130)
  Month 2 after entering the TFR phase: number analyzed (Participants) | 112 | 100
  Month 2 after entering the TFR phase | 0.1162 (0.35606) | 0.2122 (0.99372)
  Month 3 after entering the TFR phase: number analyzed (Participants) | 103 | 83
  Month 3 after entering the TFR phase | 1.3774 (9.71909) | 0.4754 (1.84649)
  Month 4 after entering the TFR phase: number analyzed (Participants) | 81 | 64
  Month 4 after entering the TFR phase | 0.2667 (0.80336) | 0.2506 (0.91197)
  Month 5 after entering the TFR phase: number analyzed (Participants) | 62 | 52
  Month 5 after entering the TFR phase | 0.1740 (0.76123) | 0.0801 (0.26739)
  Month 6 after entering the TFR phase: number analyzed (Participants) | 51 | 43
  Month 6 after entering the TFR phase | 0.2219 (1.51808) | 0.1095 (0.66322)
  Month 8 after entering the TFR phase: number analyzed (Participants) | 47 | 42
  Month 8 after entering the TFR phase | 0.0075 (0.01403) | 0.0042 (0.00742)
  Month 10 after entering the TFR phase: number analyzed (Participants) | 45 | 43
  Month 10 after entering the TFR phase | 0.0062 (0.01295) | 0.0039 (0.00680)
  Month 12 after entering the TFR phase: number analyzed (Participants) | 41 | 39
  Month 12 after entering the TFR phase | 0.0047 (0.00665) | 0.0027 (0.00357)
  Month 15 after entering the TFR phase: number analyzed (Participants) | 42 | 39
  Month 15 after entering the TFR phase | 0.0030 (0.00317) | 0.0043 (0.00555)
  Month 18 after entering the TFR phase: number analyzed (Participants) | 40 | 40
  Month 18 after entering the TFR phase | 0.0030 (0.00384) | 0.0027 (0.00330)
  Month 21 after entering the TFR phase: number analyzed (Participants) | 38 | 40
  Month 21 after entering the TFR phase | 0.0036 (0.00484) | 0.0041 (0.00495)
  Month 24 after entering the TFR phase: number analyzed (Participants) | 38 | 35
  Month 24 after entering the TFR phase | 0.0077 (0.02910) | 0.0047 (0.00691)
  Month 27 after entering the TFR phase: number analyzed (Participants) | 35 | 0
  Month 27 after entering the TFR phase | 0.0024 (0.00246) |
  Month 30 after entering the TFR phase: number analyzed (Participants) | 36 | 0
  Month 30 after entering the TFR phase | 0.0023 (0.00281) |
  Month 33 after entering the TFR phase: number analyzed (Participants) | 35 | 0
  Month 33 after entering the TFR phase | 0.0079 (0.02376) |
  Month 36 after entering the TFR phase: number analyzed (Participants) | 28 | 0
  Month 36 after entering the TFR phase | 0.0041 (0.00767) |

19. Secondary Outcome: BCR-ABL Ratio (Expressed as a Percentage) During the Nilotinib Re-treatment Phase
Description: BCR-ABL/control gene (ABL) transcript ratio by international scale (IS) (expressed as a percentage) during the nilotinib re-treatment phase. BCR-ABL is the fusion gene from breakpoint cluster region and Abelson genes.
Time Frame: From Day 1 after entering the re-treatment phase up to 24 months after entering re-treatment phase for Nilotinib 36-month treatment arm and 36 months after entering the re-treatment phase for Nilotinib 24-month treatment arm
Population: All enrolled subjects who entered the re-treatment phase. Number analyzed signified number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment Arm
Number analyzed (Participants) | 74 | 55
Percentage
  Day 1 after entering the re-treatment phase: number analyzed (Participants) | 2 | 2
  Day 1 after entering the re-treatment phase | 2.8246 (2.39596) | 0.6301 (0.74388)
  Week 6 after entering the re-treatment phase: number analyzed (Participants) | 70 | 54
  Week 6 after entering the re-treatment phase | 0.6276 (2.34231) | 0.3112 (0.60279)
  Month 3 after entering the re-treatment phase: number analyzed (Participants) | 70 | 52
  Month 3 after entering the re-treatment phase | 0.0311 (0.07265) | 0.0131 (0.02359)
  Month 6 after entering the re-treatment phase: number analyzed (Participants) | 70 | 53
  Month 6 after entering the re-treatment phase | 0.0095 (0.03296) | 0.0070 (0.01330)
  Month 9 after entering the re-treatment phase: number analyzed (Participants) | 71 | 51
  Month 9 after entering the re-treatment phase | 0.0259 (0.17766) | 0.0065 (0.01099)
  Month 12 after entering the re-treatment phase: number analyzed (Participants) | 64 | 45
  Month 12 after entering the re-treatment phase | 0.0088 (0.03190) | 0.0047 (0.00839)
  Month 15 after entering the re-treatment phase: number analyzed (Participants) | 64 | 48
  Month 15 after entering the re-treatment phase | 0.0061 (0.01322) | 0.0045 (0.01176)
  Month 18 after entering the re-treatment phase: number analyzed (Participants) | 62 | 39
  Month 18 after entering the re-treatment phase | 0.0105 (0.05205) | 0.0039 (0.00581)
  Month 21 after entering the re-treatment phase: number analyzed (Participants) | 59 | 21
  Month 21 after entering the re-treatment phase | 0.0051 (0.01699) | 0.0031 (0.00342)
  Month 24 after entering the re-treatment phase: number analyzed (Participants) | 55 | 2
  Month 24 after entering the re-treatment phase | 0.0038 (0.00756) | 0.0014 (0.00197)
  Month 27 after entering the re-treatment phase: number analyzed (Participants) | 52 | 0
  Month 27 after entering the re-treatment phase | 0.0033 (0.00439) |
  Month 30 after entering the re-treatment phase: number analyzed (Participants) | 43 | 0
  Month 30 after entering the re-treatment phase | 0.0113 (0.04446) |
  Month 33 after entering the re-treatment phase: number analyzed (Participants) | 11 | 0
  Month 33 after entering the re-treatment phase | 0.0029 (0.00541) |
  Month 36 after entering the re-treatment phase: number analyzed (Participants) | 1 | 0
  Month 36 after entering the re-treatment phase | 0.0005 (NA) — NA: Not estimable due to the low number of participants analyzed |

20. Secondary Outcome: Progression-free Survival (PFS) During the TFR Phase of the Study.
Description: PFS is defined as the time from the date of start of the nilotinib TFR phase to the date of acelerated phase/blast crisis (AP/BC) or death, whichever came first. Participants randomized in Nilotinib 36-month treatment arm had a maximum of 24 months of TFR phase, whereas participants randomized in Nilotini 24-month treatment arm had a maximum of 36 months of TFR phase.
  Patients not known to have recurred or died on or before the cut-off date for PFS analysis were censored at the date of their last assessment (cytogenetic, hematology or extramedullary) for patients who were on study, and at the date of last contact for patients who were in follow-up.
Time Frame: From the start of the TFR phase to progression to AP/BC or death up to 24 months after entering TFR phase for Nilotininb 36-month treatment arm and up to 36 months after entering TFR phase for Nilotinib 24-month treatment arm
Population: All enrolled subjects who entered the TFR phase
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment Arm
Number analyzed (Participants) | 119 | 104
Months | NA [NA to NA] — NA: Not estimable due to the low number of participants with events | NA [NA to NA] — NA: Not estimable due to the low number of participants with events

21. Secondary Outcome: Treatment -Free Survival (TFS) During the TFR Phase of the Study
Description: TFS is defined as the time from the start of the TFR phase to the date of the earliest of the following: loss of MMR, confirmed loss of MR4.0,re-start of nilotinib treatment, progression to AP/BC, or death from any cause. Patients not known to have had any of the events on or before the cut-off date were censored at the earlier of the date of their last assessment for patients who were still on study and the date of last contact for patients who were in follow-up. Participants randomized in Nilotinib 36-month treatment arm had a maximum of 24 months of TFR phase, whereas participants randomized in Nilotinib 24-month treatment arm had a maximum of 36 months of TFR phase. MMR is defined as ≥3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤0.1%BCR-ABL.
  MR4.0 is defined as either detectable disease ≤0.01%BCR-ABL IS or undetectable disease in cDNA with ≥10,000 ABL transcripts (numbers of ABL transcripts in the same volume of cDNA used to test for BCR-ABL)
Time Frame: From the start of the TFR phase to the date of occurrence of treatment-free survival event, up to 24 months after entering TFR phase for Nilotinib 36-month treatment arm and up to 36 months after entering TFR phase for Nilotinib 24-month treatment arm
Population: All enrolled subjects who entered the TFR phase
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment Arm
Number analyzed (Participants) | 119 | 104
Months | 4.1 [3.7 to 5.5] | 4.2 [3.7 to 19.7]

22. Secondary Outcome: Overall Survival (OS) Rate During the TFR Phase of the Study.
Description: OS is defined as the time from start of the TFR phase to the time of death due to any cause. Participants randomized in Nilotinib 36-month treatment arm had a maximum of 24 months of TFR phase, whereas participants randomized in Nilotini 24-month treatment arm had a maximum of 36 months of TFR phase.
  For participants without any event on or before the cut-off date, survival time will be censored at the date of their last assessment for patients who are still on study, and at the date of last contact for patients who are in follow-up.
Time Frame: From the start of the TFR phase to death due to any cause, assessed up to 24 months after entering TFR phase for Nilotinib 36-month treatment arm and up to 36 months after entering TFR phase for Nilotinib 24-month treatment arm
Population: All enrolled subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment Arm
Number analyzed (Participants) | 120 | 119
Months | NA [NA to NA] — NA: Not estimable due to the low number of participants with events | NA [NA to NA] — NA: Not estimable due to the low number of participants with events

23. Post Hoc Outcome: All Collected Deaths
Description: Deaths on-treatment were collected during the induction/consolidation phase (from the first dose of study drug to 30 days after study treatment discontinuation, assessed up to 24 months for Nilotinib 24-month treatment arm and Not randomized, and up to 36 months for Nilotinib 36-month treatment arm) and during the re-treatment phase (from the start date of the re-treatment phase to 30 days after study treatment discontinuation, assessed up to 36 months for Nilotinib 24-month treatment arm and up to 24 months for Nilotinib 36-month treatment arm).
  Total deaths were collected from first dose of study drug until end of study, up to maximum duration of 5 years
Time Frame: On-treatment deaths: induction/consolidation phase (up to 24 months or 36 months from treatment start, depending on arm) and re-treatment phase (up to 36 months or up to 24 months from re-treatment start, depending on arm). All deaths: up to 5 years
Population: All enrolled participants for whom informed consent was obtained prior to any study specific procedure were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized
Number analyzed (Participants) | 120 | 118 | 381
Participants
  On-treatment deaths | 1 | 1 | 3
  Total deaths | 1 | 3 | 10

ADVERSE EVENTS:
Time Frame: - Induction/consolidation phase: From the first dose of study drug to 30 days after study treatment discontinuation, assessed up to 24 months for Nilotinib 24-month treatment arm and Not randomized, and up to 36 months for Nilotinib 36-month treatment arm. - Re-treatment phase: From the start date of the re-treatment phase to 30 days after study treatment discontinuation, assessed up to 36 months for Nilotinib 24-month treatment arm and up to 24 months for Nilotinib 36-month treatment arm
Description: Any sign or symptom that occurred during the induction/consolidation phase and re-treatment phase. For this analysis, all enrolled participants for whom informed consent was obtained prior to any study specific procedure were included.
Groups:
- Total: Total
Arm/Group | Nilotinib 24-month Treatment | Nilotinib 36-month Treatment | Not Randomized | Total
All-Cause Mortality (participants affected / at risk) | 1/120 | 1/118 | 3/381 | 5/619
Serious Adverse Events (participants affected / at risk) | 33/120 | 27/118 | 76/381 | 136/619
Other Adverse Events (participants affected / at risk) | 97/120 | 104/118 | 280/381 | 481/619
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib 24-month Treatment (N=120) | Nilotinib 36-month Treatment (N=118) | Not Randomized (N=381) | Total (N=619)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 1 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 2 | 3
Angina pectoris (Cardiac disorders) | 0 | 0 | 5 | 5
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 4 | 9
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 4 | 4
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 3 | 3
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 4 | 6
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 2 | 3
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 2
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Death (General disorders) | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1 | 1
Hyperplasia (General disorders) | 1 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 1
Necrosis (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Sudden death (General disorders) | 0 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 3
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1 | 2
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Neuroborreliosis (Infections and infestations) | 0 | 0 | 1 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 2
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Amylase increased (Investigations) | 1 | 0 | 1 | 2
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 2 | 2
Troponin increased (Investigations) | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Cerebral artery thrombosis (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1 | 2
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 3 | 4
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 2
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 2 | 2
Mononeuropathy (Nervous system disorders) | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 2 | 4
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2 | 2
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Arterial disorder (Vascular disorders) | 0 | 0 | 1 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 1
Intermittent claudication (Vascular disorders) | 0 | 0 | 1 | 1
Ischaemia (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 2 | 3
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1 | 0 | 2
Thromboangiitis obliterans (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib 24-month Treatment (N=120) | Nilotinib 36-month Treatment (N=118) | Not Randomized (N=381) | Total (N=619)
Abdominal pain (Gastrointestinal disorders) | 7 | 6 | 15 | 28
Abdominal pain upper (Gastrointestinal disorders) | 12 | 14 | 19 | 45
Constipation (Gastrointestinal disorders) | 19 | 14 | 25 | 58
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 11 | 22
Dyspepsia (Gastrointestinal disorders) | 4 | 7 | 6 | 17
Nausea (Gastrointestinal disorders) | 13 | 5 | 11 | 29
Vomiting (Gastrointestinal disorders) | 10 | 3 | 9 | 22
Asthenia (General disorders) | 16 | 14 | 27 | 57
Fatigue (General disorders) | 13 | 7 | 17 | 37
Influenza like illness (General disorders) | 2 | 6 | 2 | 10
Pyrexia (General disorders) | 5 | 10 | 23 | 38
Bronchitis (Infections and infestations) | 8 | 9 | 14 | 31
Folliculitis (Infections and infestations) | 6 | 4 | 4 | 14
Gastroenteritis (Infections and infestations) | 10 | 3 | 4 | 17
Influenza (Infections and infestations) | 6 | 9 | 15 | 30
Nasopharyngitis (Infections and infestations) | 4 | 12 | 14 | 30
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 11 | 27
Alanine aminotransferase increased (Investigations) | 10 | 18 | 27 | 55
Aspartate aminotransferase increased (Investigations) | 8 | 12 | 11 | 31
Blood bilirubin increased (Investigations) | 8 | 13 | 30 | 51
Blood cholesterol increased (Investigations) | 15 | 14 | 24 | 53
Blood triglycerides increased (Investigations) | 3 | 8 | 6 | 17
Gamma-glutamyltransferase increased (Investigations) | 4 | 6 | 9 | 19
Lipase increased (Investigations) | 21 | 10 | 34 | 65
Weight increased (Investigations) | 5 | 6 | 3 | 14
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 5 | 12
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 7 | 5 | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 23 | 20 | 65 | 108
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 16 | 16 | 37
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 | 2 | 14 | 26
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 13 | 13 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 18 | 27 | 62
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 11 | 21 | 48
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 16 | 12 | 38
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 11 | 6 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 15 | 26 | 53
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 21 | 26 | 59
Headache (Nervous system disorders) | 17 | 12 | 34 | 63
Paraesthesia (Nervous system disorders) | 6 | 4 | 9 | 19
Sciatica (Nervous system disorders) | 5 | 7 | 9 | 21
Insomnia (Psychiatric disorders) | 4 | 6 | 3 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 15 | 13 | 37
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 9 | 18 | 33
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 15 | 17 | 41
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 23 | 57 | 95
Rash (Skin and subcutaneous tissue disorders) | 21 | 10 | 41 | 72
Hypertension (Vascular disorders) | 20 | 25 | 27 | 72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT01743989/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT01743989/SAP_001.pdf